CLINICAL TRIAL: NCT06145087
Title: Investigation of Short and Intermediate Term Effects of a Supplement Mix Designed to Target Ageing Mechanisms on Vascular Function in Healthy Middle-aged Participants (STAMINA Study)
Brief Title: Effects of a Supplement to Target Ageing Mechanisms on Vascular Function (STAMINA)
Acronym: STAMINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Principal Investigator, Prof Christian Heiss, Prof Dr, University of Surrey
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STAMINA_Protocol_V4.0
Record Dates: First submitted 2023-03-07; First posted 2023-11-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Healthy Aging; Vascular Dilation

STUDY DESIGN:
Intervention Model Description: two-armed parallel group, randomised, controlled, double-blind clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo is provided together with the placebo by AgeLess Sciences LLC, a Public Benefit Corporation.
  Interventions: Dietary Supplement: Placebo
- "NOVOS Core" supplement (Experimental): The "NOVOS Core" supplement is a commercially available product and has 12 ingredients. It was developed and is provided together with the placebo by AgeLess Sciences LLC, a Public Benefit Corporation.
  Interventions: Dietary Supplement: "NOVOS Core" supplement

INTERVENTIONS:
Dietary Supplement: "NOVOS Core" supplement — The supplement mix (15 g) is supplied as a powder to be mixed in water or other beverages like tea or coffee once per day.
  Arms: "NOVOS Core" supplement
Dietary Supplement: Placebo — The placebo mix (15 g) is supplied as a powder to be mixed in water or other beverages like tea or coffee.
  Arms: Placebo

SUMMARY:
In the ageing society, extending the healthy lifespan is a major challenge and a healthy diet may play an import role in maintaining health throughout life. With increasing age cardiovascular function declines and large and small blood vessels change in various and complex ways and these changes may lead to many age-related diseases. On a molecular level, there are many mechanisms that are associated with ageing including cellular senescence, loss of proteostasis, altered cellular communication, genomic instability, epigenetic alterations, telomere shortening, deregulated nutrient sensing, stem cell exhaustion and protein crosslinking. Animal and human studies suggest that dietary supplements may be able to affect these mechanisms. What the effect of the NOVOS Core supplement is on cardiovascular functions is not known.

The aim of the present study is to investigate the short and intermediate term effects of a supplement mix designed to target ageing mechanism on vascular function in healthy middle-aged subjects. (STAMINA Study) The hypothesis is that the supplement will lead to acute and sustained changes in biomarkers of vascular function and health.

60 healthy middle-aged people will be recruited and randomly assigned to either daily intake of the NOVOS Core supplement (n=30) or placebo (n=30) for up to 6 months (3-6). The supplement (NOVOS Core) is a commercially available product and has 12 ingredients. It was developed and is provided together with the placebo by AgeLess Sciences LLC, a Public Benefit Corporation. The study will require 2 visits by participants during which non-invasive vascular exams will be performed, venous blood taken and spot urine sample collected. The primary endpoint is change in flow-mediated dilation, secondary endpoints are change in blood pressure, cholesterol, arterial stiffness, microvascular function cardiovascular risk SCORE and daily walking distance. Tertiary endpoints are changes in biomarkers of ageing as assessed in blood samples. Measurements will be taken on the first day before and 2 hours after ingestion of the first supplement or placebo. Participants will consume the supplement or placebo for 6 months and vascular exams and one blood draw will be repeated during the final visit.

ELIGIBILITY:
Inclusion criteria:

* Generally healthy. (Note: those with stable conditions that do not interfere with the study objectives/procedures will be included at the PI discretion).
* >40 years
* Body mass index >20 kg/m2
* Systolic blood pressure >=120 mmHg
* Smartphone with step counter

Exclusion Criteria:

* Symptoms of acute infection
* Cardiac arrhythmias
* Active malignancy
* Clinical signs or symptoms of unstable cardiovascular disease (coronary artery disease, lower extremity artery disease, cerebrovascular disease). These include angina pectoris, dyspnoea, palpitation, syncope, claudication, active vasoactive medication.
* Women who have been pregnant in the last three months, currently pregnant, preparing to become pregnant during the study, or breastfeeding.
* Those that have undergone a change in hormone-based therapies such as, but not limited to, oral contraceptive pills or progesterone pills within the last 2 months. Progesterone releasing devices are considered hormone-based therapy. Spironolactone is not considered a hormone-based therapy.
* Subjects who are unwilling or unable to comply with the requirements of the protocol.
* Subjects who have a history of or a current psychological illness or condition that would interfere with their ability to understand and follow the requirements of the study in the opinion of the principal investigator.
* Subjects with or who have recently experienced traumatic injury, infections, or major surgery at the discretion of the qualified investigator.
* Subjects who are likely to start taking drugs/medication on a continuous basis or that will undergo surgery during the trial.
* Subjects engaged in donation or who were recipients of blood products within 90 days before the start of the study.
* Subjects with alcohol use of more than 2 alcoholic beverages per day within the past month.
* Subjects participated in a clinical trial with a medicinal, supplemental, nutraceutical or drug within the past two months prior to the first dose in the current study.

  * If participants take fish oil supplements, they will be asked to stop taking these supplements 21 days before the start of trial and during the trial.

Subjects using anti-inflammatory drugs on a chronic basis (e.g. aspirin, ibuprofen, diclofenac, celecoxib, etc).

* Subjects using supplements or substances present in formulation (malate, fisetin, glucosamine, alpha ketoglutaric acid, glycine, theanine, Rhodiola rosea, hyaluronic acid, ginger extract, pterostilbene, lithium). Participants will be asked to stop taking these supplements 21 days before the start of trial and during the trial.
* Subjects using supplements or substances similar as those used in the formulation (e.g. resveratrol (similar to pterostilbene) or quercetin (similar to fisetin). Participants will be asked to stop taking these supplements 21 days before the start of trial and during the trial.
* Subjects taking high-dose niacin (nicotinic acid), high-dose vitamin B3, high-dose nicotinamide (niacinamide) within 21 days before the start of the trial. Participants will be asked to stop taking these supplements 21 days before the start of trial and during the trial. .
* Subjects with clinically significant abnormal laboratory results at screening. Known allergy/intolerance to any of the components in the supplement product.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Change in flow-mediated dilation | 6 months
  Change in flow-mediated dilation with ultrasound (%)

SECONDARY OUTCOMES:
Change in systolic blood pressure | 6 months
  Change in systolic blood pressure (mmHg)
Change in diastolic blood pressure | 6 months
  Change in diastolic blood pressure (mmHg)
Change in cholesterol | 6 months
  Change in cholesterol including LDL, HDL, total cholesterol
Change in total cholesterol | 6 months
  Change in total cholesterol (mml/l)
Change in LDL cholesterol | 6 months
  Change in LDL cholesterol (mmol/l)
Change in HDL cholesterol | 6 months
  Change in HDL cholesterol (mmol/l)
Change in arterial stiffness | 6 months
  Change in pulse wave velocity (m/s)
Change in daily walking distance | 6 months
  Change in daily walking distance in kilometers as measure by personal smartphone
Change in cardiovascular risk | 6 months
  Change in calculated 10 year cardiovascular risk (European Society of Cardiology Systematic Coronary Risk Evaluation [ESC SCORE])

CONTACTS AND LOCATIONS:
Locations (1):
- University of Surrey, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT06145087/Prot_001.pdf